CLINICAL TRIAL: NCT06266221
Title: Severe Erythema Multiforme: A Randomized Controlled Trial Comparing a Short Systemic Corticosteroids Regimen to Placebo in the Acute Established Phase
Brief Title: Severe Erythema Multiforme - CORTICO
Acronym: SEMCORTICO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP200073; 2022-000712-59 (EudraCT Number)
Record Dates: First submitted 2023-05-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Erythema Multiforme
Keywords: Erythema; Corticoids; Prednisone; Methylprednisolone
MeSH Terms: conditions — Erythema Multiforme; Erythema | interventions — Prednisone; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic Corticosteroids (Experimental): Oral prednisone at 1 mg/kg/day for 3 days, tapered to 0.75 mg/kg/day for 3 days, 0.50 mg/kg/day for 3 days, 0.25 mg/kg/day for 3 days.
  If the oral route is not possible, IV methylprednisolone will be used at 0.8 mg/kg/day for 3 days, ta-pered to 0.6 mg/kg/day for 3 days, 0.4 mg/kg/day for 3 days, 0.2 mg/kg/day for 3 days (equivalent predni-sone dosage).
  In the event of a change of route administration (IV then Oral or Oral then IV), the posology of prednisone or methylprednisolone or placebo will correspond to the dosage equivalent to that prescribed at the time of the switch.
  Interventions: Drug: Prednisone 20 Mg; Drug: Methylprednisolone 120 Mg
- Placebo (Placebo Comparator): Oral or IV placebo with the same decrease of dose: same number of tablets for prednisone placebo and same volume as methylprednisolone for its placebo
  Interventions: Drug: Oral Placebo; Drug: IV Placebo

INTERVENTIONS:
Drug: Prednisone 20 Mg — Oral corticosteriods
  Other Names: Oral corticosteriods
  Arms: Systemic Corticosteroids
Drug: Oral Placebo — Oral placebo
  Other Names: placebo
  Arms: Placebo
Drug: Methylprednisolone 120 Mg — IV corticosteriods
  Other Names: IV corticosteriods
  Arms: Systemic Corticosteroids
Drug: IV Placebo — IV placebo
  Other Names: placebo
  Arms: Placebo

SUMMARY:
Erythema multiforme (EM) is an acute and often recurrent mucocutaneous disease. EM is considered a hypersensitivity immune-mediated reaction. The two main known triggering factors are Herpes simplex virus (HSV) and Mycoplasma pneumoniae (MP) infections. Typical target skin lesions characterize EM, especially oral MMs. EM is in fact mainly linked to the oral MM involvement, including intense mucosal pain, impaired food intake, weight loss, hospitalization and potential risk of fibrotic sequelae (oral, ocular, genital, oesophageal, respiratory tract) and recurrences.

The objectives of treatment for severe EM in the acute phase are to reduce the duration of lesions, prevent complications and mucosal sequelae. However, despite the lack of evidence and consensus some medical teams often use a short regimen of SCS hoping to obtain a quicker improvement of the condition. However, the use of SCS at the acute phase is not codified and remains debated according to the existent literature. Current studies are mostly retrospective and based on small cohorts or case reports. A randomized, controlled trial would be therefore essential to properly evaluate the benefit of SCS in this pathology and provide strong support to clinicians in their decision making in severe EM during the acute phase.

This research will be a Phase III randomized, multicentric, double-blind, controlled trial with two parallel groups. The efficacy of prednisone, oral at 1 mg/kg/day for 3 days, tapered to 0.75 mg/kg/day for 3 days, 0.50 mg/kg/day for 3 days, 0.25 mg/kg/day for 3 days is compared to that of placebo, oral for 12 days or IV methylprednisolone if oral route is impossible because of the self-reported inability for the patient to swallow due to the impacts of the oral lesions, with dosage equivalence at 0.8 mg/kg/day for 3 days, tapered to 0.6 mg/kg/day for 3 days, 0.4 mg/kg/day for 3 days, 0.2 mg/kg/day for 3 days, then stopped, compared to that of placebo.

A stratification according to the food intake classification (0,1,2 vs 3) will be performed.

An interim analysis is planned after the inclusion of 50 patients. Results of the interim analysis will be presented to the DSMB. During the interim analysis, inclusions may continue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 15 years old and 30 kg ≤ Weight ≤ 150 kg
* Clinical diagnosis of severe EM defined as:

  * Typical skin lesions if first flare of EM: raised target lesions with 2 or 3 concentric rings located on the extremities or disseminated. In case of recurrent EM, with proven anterior flare (known clinical diagnosis as-sociating typical skin lesions and MM involvement in a previous flare), typical skin lesions are not essential for inclusion, because EM may manifest as isolated mucosal involvement.
  * Two or more MMs affected (mouth, throat, eyes, ear, nose, genital and/or anal areas), or only the oral MM affected, if severely affected (score* 2 or 3 of Harman criteria22) with altered general conditions and significant impact on food intake (solid food impossible)
* First flare of EM or acute recurrence of previously diagnosed EM
* Disease flare that has lasted for up to 5 days (≤5 days)
* Affiliated to a social security scheme
* Able to provide written informed consent; consent of both parents will be col-lected for minors

  * score: 1, minor activity (up to three erosions); 2, moderate activity (more than three but less than 10 erosions, or generalized desquamative gingivitis); 3, severe (more than 10 discrete erosions or extensive, confluent erosions, or generalized desquamative gingivi-tis with discrete erosions at other oral sites).

Exclusion Criteria:

* EM without involvement of oral cavity compromising normal solid food
* Patients unable to eat solid food outside of their current pathology (erythema multiforme)
* Other diagnosis potentially involving MMs: Stevens-Johnson syndrome and toxic epidermal necrolysis (SJS/TEN), pemphigus, herpetic gingivostomatitis
* Systemic Corticosteroids prescribed for another disease on inclusion day (any dose)
* Use of systemic Corticosteroids for > 5 days for any previous flare of EM (>10mg),
* Contraindication to systemic Corticosteroids:

  * hypersensitivity to systemic Corticosteroids or to an excipient;
  * uncontrolled primary bacterial, viral, fungal or parasitic infection
  * psychotic states not yet controlled by treatment
* Sepsis (shock, cyanosis, hypothermia, low blood pressure monitored succes-sively twice (systemic blood pressure < 90 mmHg and diastolic blood pres-sure < 60 mmHg)
* Kidney or liver insufficiency (creatinine level ≥ 150 µmol/L; aspartate ami-notransferase or alanine aminotransferase level > 3 times the upper limit of normal)
* Current cancer with the exception of non-metastatic skin carcinoma not re-quiring immediate medical treatment
* Pregnant or breastfeeding
* Person subject to safeguards of justice
* Person deprived of liberty by judicial or administrative decision
* Person subject to psychiatric care without their consent
* Person admitted to a health or social establishment for purposes other than those of research
* Person unable to express their consent
* Person under legal protection (guardianship or curatorship)
* Participation in another interventional study involving human participants or in the exclusion period at the end of a previous study involving human partici-pants, if applicable
* On state medical aid

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Time to success | Day0 to Month1
  It will be defined by controlled pain (Numeric Rating Scale (NR, range 0-10) score <4 and sustained no need for any level III analgesics, during 48 hours), resumption of non-blended food intake and no need for rescue therapy (IV methylprednisolone at 1mg/kg/day with discontinuation of the current treatment in both arms).
Evaluation of Pain | Day0 to Month1
  It will be evaluated daily by using the NR (0-10), 3 times a day during hospitalization and once a day (worst score of the day) after the hospitalization by phone until achievement of the primary end-point. To avoid confounding bias, management of pain will be standardized: Level I, II and III analgesics will be permitted during the treatment, but analgesics taken will be reported and the success is defined as no need for any level III analgesics.
Food intake | Day0 to Month1
  It will be evaluated qualitatively daily by the investigator team (eg. investigator or collaborator, dietician, trained clinical study technician) by use of a standardized questionnaire. Food intake will be classified as the following categories: 0, impossible to eat; 1, liquid food possible; 2, mixed food possible; 3, chopped food possible; 4, solid food possible. For patient with categories 0, 1 or 2 at baseline, the success will be defined by the resump-tion of categories 3 or 4. For patients with category 3 at baseline, the success will be catego-ry 4.
  A subgroup analysis will be performed considering the two food intake classification strata.
Rescue therapy intake | From Day 0 until discharge from hospital, assessed up to Day 15
  The rescue therapy will be standardized for all patients in failure of the initial strategy and will be:
  IV methylprednisolone at 1 mg/kg/day with discontinuation of the current treatment in both arms.

SECONDARY OUTCOMES:
Time to clear or almost clear healing of all sites | Day15 and Month1
  "clear" is defined as no erosion or skin ulceration and absence of new lesions and "almost clear" is defined as "presence of 1, or 2 maximum, micro erosions / punctiform millimetric erosions, and absence of new lesions". Healing will be evaluated by the clinician. To avoid bias, the investigators will be trained before the start of the study allowing a standardization of the evaluation of healing
Time to fever resolution | From Day 0 until discharge from hospital, assessed up to Day 15
  fever resolution defined as absence of fever (temperature ≤ 37,8°C) for at least 24 h
Length of hospital stay | From Day 0 until discharge from hospital, assessed up to Day 15
Number of days of consumption of level III analgesics | From Day 0 until complete healing, assessed up to Month 1
  at least once in the day
Evaluation of pain | From Day 0 until complete healing, assessed up to Month 1
  It will be assessed three times a day during hospitalization and once a day (worst score of the day) after the hospitalization until achievement of the primary endpoint.
Chopped or solid food intake resumption | From Day 0 until complete healing, assessed up to Month
Rate of patients in the two groups with need for a rescue therapy | From Day 0 until discharge from hospital, assessed up to Day 15
  The rescue therapy will be standardized for all patients in failure of the initial strategy and will be:
  IV methylprednisolone at 1 mg/kg/day with discontinuation of the current treatment in both arms.
Rate of sequelae | Month3 and Month6
  cutaneous and mucosal sequelae (ocular, ENT, esophageal, pulmonary and genital sequelae)), assessed clinically at month 3 (M3, if realized) and month 6 (M6)
Rate of adverse events during the treatment and follow-up | Day0 to Month6
Evaluation of the quality of life | at the end of hospitalization, Day7, Day15 and Month1 and in case of relapse
  It will be performed with the use of Patient Global Impression of Change (PGIC), scale on 7 points

CONTACTS AND LOCATIONS:
Overall Officials: Candy Estevez, M.Sc, Study Chair — APHP

IPD SHARING:
Plan to Share IPD: No